CLINICAL TRIAL: NCT03320954
Title: Language Assessment and Treatment Following Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17512
Record Dates: First submitted 2017-10-09; First posted 2017-10-25 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Brain Injuries
Keywords: Language; Anomia
MeSH Terms: conditions — Brain Injuries; Language; Anomia

STUDY DESIGN:
Intervention Model Description: Phase 1 participants will include people with and without acquired brain injuries. This phase does not involve any intervention.
  Phase 2 participants will include only people with acquired brain injuries. This portion of the research involves an intervention procedure. All participants will receive the same intervention.
  Phase 3 participants will be limited to those people with acquired brain injuries who completed Phases 1 and 2. Phase 3 does not involved any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anomia treatment (Experimental): Phase 2 portion of the research during which participants with acquired brain injury will perform intervention activities.
  Interventions: Behavioral: Anomia treatment

INTERVENTIONS:
Behavioral: Anomia treatment — Phase II participants will attend two-hour, group intervention sessions one day per week for eight weeks. Participants will engage in multiple word game activities throughout each intervention session. Games will include Facts in Five, Anomia, Boggle, and Bananagrams as well as variations on these, as appropriate.

SUMMARY:
People with acquired brain injury (ABI) often experience persistent language challenges that are subtle in nature and not readily observable to others. These challenges can have substantial negative effects on vocational and social endeavors despite their subtlety. Even though these challenges are prevalent in the ABI population, limited methods exist for quantifying and remediating them. The two purposes of Phase I of this research are to (a) explore methods of using event related potential (ERP) recordings to quantify language processing differences between people with and without ABI and (b) correlate behavioral observations from language tests with ERP findings. The purpose of Phase II is to explore the use of game-based, group activities as an intervention for people with ABI who experience word-retrieval challenges. The purpose of Phase III is to collect post-intervention data for comparison with Phase I data and provide evidence about the effectiveness of the intervention program.

DETAILED DESCRIPTION:
Phase I: Phase I participants will engage in two sets of activities: (a) standardized and informal language and cognitive measures and (b) a series of language and cognitive activities performed during the collection of event related potential (ERP) recordings. Standardized language measures will include the: (a) Test of Adolescent/Adult Word Retrieval, (b) Cognitive Linguistic Quick Test, and (c) California Verbal Learning Test. Informal measures will include a conversational interaction about a participant's language difficulties and a topic of his/her choosing. During the conversational interaction, participants will press a button each time they experience difficulty retrieving a word.

ERPs measure electrical signals from the brain using a soft net of woven electrodes placed on a participant's head. Before the session, the investigators will soak a net in a saline (salt water) solution. The recording electrodes will be placed on the participant's scalp. The investigators will record ERPs while the participant completes the following tasks:

1. word retrieval: The participant will view a series of neutral stimuli (i.e., pictures of familiar objects, people, or locations flashed briefly on a computer monitor). The participant will press one of three buttons to indicate (a) recall of the name of the depicted image, (b) knowledge of the name but inability to recall it, or (c) no knowledge of the name of the depicted image. If a participant does not press a button within the time limit of the stimulus presentation, a new stimulus trial will begin. During some trials, participants will perform a second task requiring judgment about the orientation of lines appearing after the stimulus image. Following completion of all trials, the investigators will present the stimulus images a second time along with three response options: (a) the correct name, (b) an incorrect name, and (c) "don't know." The participant will again use a button press to indicate his/her response choice.
2. stimulus categorization: The participant will view a series of objects. For each object, he/she will categorize the stimulus semantically (e.g., Is the object a fruit or animal?) or phonologically (e.g., Does the object start with the letter "L" or "N?"). Participants will respond by pushing a button.
3. deductive reasoning: The participant will view written word pairs. Some of the pairs will relate to a specific word (e.g., "desert" and "humps" relate to "camel"), whereas other pairs will not (e.g., "desert" and "bark"). The participant will press one of two buttons to indicate whether a word pair triggers or does not trigger recall of a related word.

Phase II: Only people with acquired brain injury (ABI) will participate in Phase II activities. Phase II participants will attend two-hour, group intervention sessions one day per week for eight weeks. Participants will engage in multiple word game activities throughout each intervention session. Games will include Facts in Five, Anomia, Boggle, and Bananagrams as well as variations on these, as appropriate. Data collection during these sessions will be limited to a list of activities in which a participant engaged and the duration of engagement in each activity. Game-based group activities such as these are not typically used in intervention sessions for people with ABI who experience mild word-retrieval challenges. In fact, because of the subtlety of word retrieval difficulties experienced by people with relatively good recoveries from ABI--that is, the target population for this research--most people do not receive any treatment for this problem.

Phase III: Only people with ABI who have performed both Phase I and Phase II activities will be eligible for participation in Phase III. Following completion of the intervention sessions, participants will perform post-testing activities. Post-testing activities will include a subset of Phase I testing activities. Specifically, we will repeat (a) the audio recording of a conversational interaction and (b) the ERP recording with the same tasks used in Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Adults with acquired brain injury (ABI):
* Have sustained a mild, moderate, or severe ABI
* Have concerns about language-related challenges following ABI
* Adults without ABI
* Have no history of ABI, other neurological impairment, or learning challenges
* Match a participant with ABI on age, gender, and education

Exclusion Criteria:

* Do not speak English as a primary language

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Change in amplitude of N400 event related potential (ERP) as measured in microvolts. | The second day of participant enrollment and 10 weeks later on the last day of participant enrollment
  ERP recordings will be taken while a participant performs naming tasks. The average amplitude of N400 will be measured in microvolts across trials.

SECONDARY OUTCOMES:
Total raw score on Test of Adolescent/Adult Word Retrieval | First day of participant enrollment
  A participant will perform the Test of Adolescent/Adult Word Retrieval. Scoring will be done in accordance with the standardized procedures outlined in the manual. Possible scores range from 0-107, with higher scores indicating better performance than lower scores.
Executive Functions Domain score on the Cognitive Linguistic Quick Test | First day of participant enrollment
  A participant will perform the Cognitive Linguistic Quick Test. Scoring will be done in accordance with the standardized procedures outlined in the manual. Executive Functions Domain scores are the sum of the scores obtained on the Symbol Trails task (range: 0-10), the Generative Naming task (range: 0-9), the Mazes task (range: 0-8), and the Design Generation task (range: 0-13). Possible Executive Function Domain scores range from 0 to 40, with higher scores indicating better performance than lower scores. Scores from 0-15 correspond with a severity rating of 1; scores from 16-19 correspond with a severity rating of 2; scores from 20-23 correspond with a severity rating of 3; and scores from 24-40 correspond with a severity rating of 4 and performance within normal limits.
Visuospatial Domain score on the Cognitive Linguistic Quick Test | First day of participant enrollment
  A participant will perform the Cognitive Linguistic Quick Test. Scoring will be done in accordance with the standardized procedures outlined in the manual. Visuospatial Domain scores are the sum of the scores obtained on the Symbol Cancellation task (range: 0-12) times 2, the Symbol Trails task (range: 0-10) times 2, the Design Memory task (range: 0-6) times 4, the Mazes task (range: 0-8) times 3, and the Design Generation task (range: 0-13) times 1. Possible Visuospatial Domain scores range from 0 to 105, with higher scores indicating better performance than lower scores. Scores from 0-41 correspond with a severity rating of 1; scores from 42-51 correspond with a severity rating of 2; scores from 52-81 correspond with a severity rating of 3; and scores from 82-105 correspond with a severity rating of 4 and performance within normal limits.
Trials 1-5 Free Recall Total Correct on the California Verbal Learning Test - II | First day of participant enrollment
  A participant will perform the California Verbal Learning Test. Scoring will be done in accordance with the standardized procedures outlined in the manual. Raw scores range from 0 to 100. Higher total correct scores indicate better performance than lower total correct scores.
Change in number of self-reported instances of word retrieval difficulty | The second day of participant enrollment and 10 weeks later on the last day of participant enrollment
  A participant will engage in a conversational interaction with the researcher. The participant will press a button each time he/she experiences difficulty retrieving a word. The number of instances of self-reported word retrieval difficulty will be tallied.
Amplitude of N400 event related potential (ERP) as measured in microvolts. | First day of participant enrollment
  ERP recordings will be taken while a participant performs naming tasks. The average amplitude of N400 will be measured in microvolts across trials.

OTHER OUTCOMES:
Time spent performing specific intervention activities | Weeks two through nine of participant enrollment
  The investigators will measure the amount of time each participant chooses to spend engaging in specific game activities during the Phase II intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Hux, PhD, Principal Investigator — University of Nebraska Lincoln; Kathy Chiou, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share IPD data because they do not believe the data can be adequately de-identified to protect the privacy of participants. This is because individuals with ABI constitute a relatively small number of people within the local community.